CLINICAL TRIAL: NCT04748991
Title: Vernakalant Versus Amiodarone for Post-operative Atrial Fibrillation in Cardiac Surgery Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB20-2257
Record Dates: First submitted 2021-01-25; First posted 2021-02-10 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Post-cardiac Surgery
Keywords: Amiodarone; Vernakalant
MeSH Terms: conditions — Atrial Fibrillation | interventions — vernakalant; Amiodarone

STUDY DESIGN:
Intervention Model Description: Patients will be recruited from the CVICU 24 hours after admission to CIVCU based on inclusion and exclusion criteria. Patients identified with new presentation atrial fibrillation with a sustained duration of greater than 30 minutes will be considered for the study. Patients will be randomized to Amiodarone versus Vernakalant using a computerized process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Vernakalant (Experimental): Patients randomized to Vernakalant will receive a bolus of 3mg/kg over 10 minutes and an observation period of 15 minutes, if the patient is still in AF, they will receive an additional 2.0mg/kg bolus of Vernakalant.
  Interventions: Drug: Vernakalant
- Intravenous Amiodarone (Active Comparator): Patients randomized to an amiodarone arm will receive 150mg IV bolus and an amiodarone infusion of 1mg/hr x 6 hours followed by 0.5mg/hr x 12 hours.
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Vernakalant — Post operative AF after cardiac surgery. Vernakalant 3mg/kg over 10 minutes followed by 2mg/kg over 10 minutes if still in AF.
  Other Names: BRINAVESS
  Arms: Intravenous Vernakalant
Drug: Amiodarone — Post operative AF after cardiac surgery. Amiodarone 150mg IV followed by 1 mg/min x 6 hours then 0.5 mg/min x 12 hours
  Other Names: Cordarone, Nexterone, Pacerone
  Arms: Intravenous Amiodarone

SUMMARY:
Post-operative atrial fibrillation is a common problem post cardiac surgery with rates exceeding 30%. Atrial fibrillation has multiple adverse effects on cardiac hemodynamics and can lead to hypotension, diminished end organ perfusion and lengthen the stay in ICU. Amiodarone is the medication of choice used for pharmacological cardioversion and can be used with vasoactive medications. Intravenous amiodarone is associated with hypotension and end organ perfusion requiring escalation in vasoactive support. Vernakalant is novel anti-arrhythmic agent approved in Canada for cardioversion of atrial fibrillation that primarily works on atrial channels and has no effect on contractility or vasodilation. Clinical trials have proved good efficacy of Vernakalant in conversion of paroxysmal atrial fibrillation however there is no comparison of Amiodarone to Vernakalant in post-operative cardiac surgery. We plan to perform a clinical trial comparing Vernakalant to amiodarone in post-cardiac surgery patients with a primary outcome of cardioversion at 90 minutes. Secondary outcomes will follow duration of vasoactive medications, days in ICU and economics.

DETAILED DESCRIPTION:
1. Background - Atrial fibrillation (AF) is the most common cardiac arrhythmia post cardiac surgery. Estimates suggest that rates of patients experiencing post-operative atrial fibrillation (POAF) after cardiac surgery exceeds 30%. Atrial fibrillation has multiple effects on the cardiopulmonary hemodynamics. Rapid irregular ventricular rate results in decreased coronary flow diminishing the ability to preserve myocardial oxygen demand leading to ischemia. Atrial contraction provides 15-20% of LV filling in normal cardiac physiology and loss of synchronized atrial contraction in addition to decreased diastolic filling time may lead to decreased cardiac. This may lead to hypotension and diminished end organ perfusion requiring additional vasoactive support. Currently amiodarone is utilized as the pharmacological agent of choice for POAF in cardiac surgery, typical rate control agents are contraindicated due to need of vasoactive requirements. However direct effects of IV amiodarone include vasodilation and hypotension typically requiring escalating doses of vasoactive medications, which subsequently prolong stay in the CVICU (cardiovascular Intensive Care Unit), increase exposure to vasopressors and potentially mechanical ventilation. Vernakalant is a Von Williams Class III novel anti-arrhythmic agent with primary activity on atrial tissue with limited activity on ventricular myocardium. Primary mechanism of action is blocking early activating K+ atrial channels and frequency-dependent atrial Na+ channels which prolongs atrial refractory periods and decreasing atrial conduction without promoting ventricular arrhythmia. There have been many trials that proven efficacy in converting AF in patients with atrial fibrillation and in the post cardiac surgery patients, however this has never been compared to standard of care Amiodarone.
2. Research Questions and objectives: We hypothesize administration of vernakalant compared to amiodarone will have a higher rate of cardioversion to sinus rhythm at 90 min in post-operative sustained atrial fibrillation. This will reduce duration of vasoactive medications, days in ICU and mortality.
3. Methods: Patients will be recruited from the CVICU 24 hours after admission to CIVCU based on inclusion and exclusion criteria. Patients identified with new presentation atrial fibrillation with a sustained duration of greater than 30 minutes will be considered for the study. Patients will be randomized to Amiodarone versus Vernakalant using a computerized process. Patients randomized to an amiodarone arm will receive 150mg IV bolus and an amiodarone infusion of 1mg/hr x 6 hours followed by 0.5mg/hr x 12 hours. Patients randomized to Vernakalant will receive a bolus of 3mg/kg over 10 minutes and an observation period of 15 minutes, if the patient is still in AF, they will receive an additional 2.0mg/kg bolus of Vernakalant. Infusions will be discontinued if QT interval becomes >550ms, heart rate less than 45 bpm lasting >30 seconds with symptoms or <40bpm lasting >30 seconds with or without symptoms, ventricular tachycardia or development of heart block. At 90 minutes rate of conversion to sinus rhythm will be documented. Secondary outcomes including time to AF conversion, recurrence of atrial fibrillation will be documented along with safety events over 48h. Duration of vasoactive medications, days in ICU, time to initiation of beta blockers, mortality, Left Ventricular (LV) function and economics of ICU still will be followed. Patients will be excluded if they return to the OR.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/=18 years
2. Undergone heart surgery for coronary artery bypass surgery (on-pump or off-pump CABG) and/or valve repair or replacement (excluding mechanical valves), including re-operations.
3. Hemodynamically stable with/without vasopressor support

Exclusion Criteria:

1. LVAD insertion or heart transplantation
2. MAZE procedure
3. Transcatheter aortic valve replacement (TAVR)
4. History of or planned mechanical valve replacement
5. Rheumatic heart disease
6. Congenital cardiac defect (excluding bicuspid aortic valve or patent foramen ovale)
7. History of prior atrial fibrillation or flutter
8. History of ablation for atrial fibrillation
9. Contraindication to amiodarone

   * PR >240ms
   * Heart block (2nd or 3rd degree)
   * QTC >480ms
   * Untreated thyroid disorder
   * AST or ALT >2x upper limit of normal
   * Hepatic cirrhosis
   * Interstitial lung disease
10. Received amiodarone within 6 weeks
11. Contraindications to Vernakalant

    * Known hypersensitivity to Vernakalant
    * Prolonged QT
    * Heart block (2nd or 3rd degree)
    * Use of anti-arrhythmic medication in the past 4 weeks.
12. Return to OR during CVICU stay or readmission to CIVCU from Cardiac Surgery ward.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Rate of conversion of sustained post-operative atrial fibrillation at 90 minutes. | 90 minutes
  Rate of conversion of sustained post-operative atrial fibrillation at 90 minutes.

SECONDARY OUTCOMES:
Duration of vasopressor therapy | 7 days
  Duration of vasopressor therapy
Time to conversion to sinus rhythm | 7 days
  Time to conversion to sinus rhythm
Days in intensive care unit | 7 Days
  Days in intensive care unit
Recurrence of atrial fibrillation within 48 hours | 48 hours
  Recurrence of atrial fibrillation within 48 hours
Mortality | 1 month
  Mortality
LV function (Normal, Mild, Moderate or Severe) | 7 days
  LV function (Normal, Mild, Moderate or Severe)
Time to initiation of beta-blockers | 7 days
  Time to initiation of beta-blockers
Economics - cost of hospital stay | Up to one month
  Economics - cost of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chiu, MD, MSC, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roy D, Pratt CM, Torp-Pedersen C, Wyse DG, Toft E, Juul-Moller S, Nielsen T, Rasmussen SL, Stiell IG, Coutu B, Ip JH, Pritchett EL, Camm AJ; Atrial Arrhythmia Conversion Trial Investigators. Vernakalant hydrochloride for rapid conversion of atrial fibrillation: a phase 3, randomized, placebo-controlled trial. Circulation. 2008 Mar 25;117(12):1518-25. doi: 10.1161/CIRCULATIONAHA.107.723866. Epub 2008 Mar 10. PMID 18332267
- [Background] Kowey PR, Dorian P, Mitchell LB, Pratt CM, Roy D, Schwartz PJ, Sadowski J, Sobczyk D, Bochenek A, Toft E; Atrial Arrhythmia Conversion Trial Investigators. Vernakalant hydrochloride for the rapid conversion of atrial fibrillation after cardiac surgery: a randomized, double-blind, placebo-controlled trial. Circ Arrhythm Electrophysiol. 2009 Dec;2(6):652-9. doi: 10.1161/CIRCEP.109.870204. PMID 19948506
- [Background] Camm AJ, Capucci A, Hohnloser SH, Torp-Pedersen C, Van Gelder IC, Mangal B, Beatch G; AVRO Investigators. A randomized active-controlled study comparing the efficacy and safety of vernakalant to amiodarone in recent-onset atrial fibrillation. J Am Coll Cardiol. 2011 Jan 18;57(3):313-21. doi: 10.1016/j.jacc.2010.07.046. PMID 21232669
- Available data/document: Product monograph - Vernakalant — https://pdf.hres.ca/dpd_pm/00038441.PDF
- Available data/document: Product monograph - Amiodarone — https://pdf.hres.ca/dpd_pm/00035425.PDF